CLINICAL TRIAL: NCT05289648
Title: The Molecular and the Clinical Effects of Preoperative Niraparib in Patients with High-grade Endometrial Cancer: Phase 0 Exploratory Trial
Brief Title: Niraparib in High-grade Endometrial Cancer Trial
Acronym: NIREC
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to obtain funding
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Shannon Salvador, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 301014
Record Dates: First submitted 2022-02-18; First posted 2022-03-21 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer; Serous Adenocarcinoma; Uterine Neoplasm
Keywords: Biomarker; Chemotherapy naïve; Synthetic lethality; Phase 0
MeSH Terms: conditions — Endometrial Neoplasms; Cystadenocarcinoma, Serous; Uterine Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preoperative Niraparib (Experimental): Single arm. Following the initial assessment and endometrial biopsy the participants will receive niraparib for 28 days. After the treatment period the patients will be surgically staged. All participants will receive the standard of care.
  Interventions: Drug: Niraparib oral capsule

INTERVENTIONS:
Drug: Niraparib oral capsule — Low dose oral niraparib capsules (2 x 100 mg) once a day for 28 days
  Other Names: Zejula

SUMMARY:
The study will investigate the effect of niraparib on tumor tissue in chemotherapy naïve, newly diagnosed, high-grade endometrial cancer patients. Biomarkers of cognate molecular pathways as well as investigational assays will be used to study the antineoplastic effect of the drug.

DETAILED DESCRIPTION:
Niraparib is a FDA approved Poly(ADP-ribose) polymerase inhibitor (PARPi) for the treatment of platinum-sensitive ovarian serous carcinoma. The safety profile of niraparib was established in phase III clinical trials. The therapeutic effect of niraparib on serous endometrial carcinoma is now being investigated in several clinical trials. However, the antineoplastic effect and the safety profile of niraparib in chemotherapy naïve high-grade endometrial cancer patients is unknown. By employing a phase 0 exploratory trial design, the investigators will study the niraparib's effect on endometrial cancer in chemotherapy naïve patients using molecular biomarkers as sentinels for the antineoplastic effect. Women diagnosed by endometrial biopsy with high-grade endometrial cancer will receive niraparib for 28 days. Staging surgery will be performed 4-6 weeks after the diagnosis (standard of care). The investigators will use the pre-operative biopsy and the surgical specimen to perform comparative multidimensional analysis of endometrial tumors before and after exposure to niraparib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female ≥18 years of age, able to understand the study procedures and agree to participate in the study by providing written informed consent
2. Histological and staging criteria:

   Patients must have histologically diagnosed
   1. Grade 3 endometrioid, serous or clear cell endometrial carcinoma, carcinosarcoma, undifferentiated carcinoma in Stage I-III according to International Federation of Gynecology and Obstetrics (FIGO) classification.
   2. Grade 2 endometrioid carcinoma with abnormal TP53 by immunohistochemistry.
3. Surgical criteria: patients with operable disease are eligible
4. Patients of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin [hCG]) within 7 days prior to receiving the first dose of niraparib.
5. Patients must be postmenopausal, free from menses for >1 year, surgically sterilized, or willing to use adequate contraception to prevent pregnancy or must agree to abstain from activities that could result in pregnancy throughout the study, starting with enrollment through 3 months after the last dose of niraparib.
6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Patients must have adequate organ function, defined as follows:

   1. Absolute neutrophil count ≥ 1,500/µL
   2. Platelets ≥ 100,000/µL
   3. Hemoglobin ≥ 10 g/dL
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault equation
   5. Total bilirubin ≤ 1.5 x ULN
   6. Aspartate aminotransferase and alanine aminotransferase ≤ 2.0 x ULN
8. Patients must be able to take oral medications

Exclusion Criteria:

1. Histology:

   1. Grade 1 endometrioid carcinoma OR
   2. Grade 2 endometrioid carcinoma with wild type TP53 OR
   3. Grade 2 endometrioid carcinoma with an unknown TP53 status
2. Patient did not consent for the study biopsy and one of the following:

   * the original endometrial biopsy tissue block could not be assessed by the study site pathologist
   * the original endometrial biopsy tissue block does not contain sufficient tumor tissue
3. Patient is pregnant, breastfeeding, or expecting to conceive children, while receiving study treatment and for 3 months after the last dose of study treatment;
4. Patient has a known hypersensitivity to the components of niraparib or its excipients;
5. Patient is simultaneously enrolled in any clinical trial of niraparib or any other investigational therapy;
6. Patient has had any known ≥Grade 3 anemia, neutropenia or thrombocytopenia due to any prior medication that persisted >4 weeks;
7. Patient has any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myelocytic anemia (AML);
8. Patient has undergone major surgery (per investigator judgment) within 3 weeks of starting the study or patient has not recovered from any effects of any major surgery;
9. Patient has a condition (such as transfusion dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results or interfere with the patient's participation for the full duration of the study treatment, including:

   1. Patient received a transfusion (platelets or red blood cells) within 2 weeks of the first dose of study treatment;
   2. Patient received colony-stimulating factors (eg, granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 2 weeks prior to the first dose of study treatment.
10. Another concurrent invasive neoplastic disease (including ovarian), diagnosis of cancer in the last 5 years (except for non-melanoma skin cancer), patient previously had cancer (> 5 years) but she is not considered cured or still treated.
11. Patient is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection;

    - Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
12. Patient is immunocompromised (patients with splenectomy are allowed).
13. Patient has known, active hepatic disease (ie, hepatitis B or C).
14. Patient has a corrected QT interval (QTc) prolongation > 470 milliseconds at screening; - If a patient has a prolonged QTc interval and the prolongation is deemed to be due to a pacemaker upon investigator evaluation (ie, the patient otherwise has no cardiac abnormalities), then the patient may be eligible to participate in the study following approval of a cardiology specialist.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Tumor cells proliferation before and after the treatment | Day 30 (day of surgery)
  Cancer cell proliferation will be quantitatively assessed using immunohistochemical staining for cell-cycle proteins.
  Ki-67 (MIB) stains nuclei of cells in G1-S-G2 phases of the cell-cycle. The proliferation index will be calculated as percent of tumor positive cells. The primary outcome fold change in proliferation index after exposure to niraparib. The quantification will be done by image analysis software with pathologist supervision.
Cell cycle arrest | Day 30 (day of surgery)
  The levels of different cell-cycle related proteins increase and decrease throughout the cell cycle, each having its own expression pattern.
  Tumor specimens will be stained for Cyclin D1, Geminin and p21 proteins. The proportion of positive nuclei of each marker after exposure to niraparib will be estimated. The results will be integrated to study the effect of niraparib on endometrial cancer cells proliferation.
Apoptosis marker | Day 30 (day of surgery)
  Cleaved caspase-3 (cCas-3) marks cells that activated the programmed cell-death process. cCas-3 positive tumor cells will be compared before and after the exposure to niraparib.

SECONDARY OUTCOMES:
Endometrial thickness | Day 1 and Day 28
  Comparison of the thickness of endometrial lining before and after treatment
CA-125 cancer tumor marker | Day 1 and Day 28
  Investigation of the effect of preoperative niraparib on CA125 levels in patients with high grade endometrial carcinoma
Adverse effects of Niraparib | every week from day 1 and 21 days after the surgery
  Assessment of adverse effects of niraparib in chemotherapy naïve patients according to CTCAE 5.0
Patient Reported Outcomes - General Oncology | Day 1 and Day 28
  Patients' well being will be assessed by a validated questionnaire: Functional Assessment of Cancer Therapy - General (FACT-G). https://www.facit.org
Patient Reported Outcomes - Endometrial Cancer | Day 1 and Day 28
  Patients' well being will be assessed by a validated questionnaire: Functional Assessment of Cancer Therapy - Endometrial (FACT-en). https://www.facit.org

OTHER OUTCOMES:
Alternation in genes expression | Day 30 (day of surgery)
  Gene expression profile by RNA sequencing extracted from snap-frozen tumor tissue. Unsupervised hierarchical clustering of 2-fold changed genes will be used to detect the pathways affected by niraparib treatment.
Genomic analysis | Day 30 (day of surgery)
  Mutational signature and the altered genes of the DNA repair pathway will be identified by DNA next generation sequencing. Genomic findings will be correlated with molecular analysis for discovery of biomarkers for niraparib sensitivity in chemotherapy-naïve endometrial cells.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Salvador, MD MSc, Principal Investigator — McGill University, Jewish General Hospital; Walter Gotlieb, MD PhD, Principal Investigator — McGill University, Jewish General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Jonge MM, Auguste A, van Wijk LM, Schouten PC, Meijers M, Ter Haar NT, Smit VTHBM, Nout RA, Glaire MA, Church DN, Vrieling H, Job B, Boursin Y, de Kroon CD, Rouleau E, Leary A, Vreeswijk MPG, Bosse T. Frequent Homologous Recombination Deficiency in High-grade Endometrial Carcinomas. Clin Cancer Res. 2019 Feb 1;25(3):1087-1097. doi: 10.1158/1078-0432.CCR-18-1443. Epub 2018 Nov 9. PMID 30413523
- [Background] Urick ME, Bell DW. Clinical actionability of molecular targets in endometrial cancer. Nat Rev Cancer. 2019 Sep;19(9):510-521. doi: 10.1038/s41568-019-0177-x. Epub 2019 Aug 6. PMID 31388127
- [Background] Mirza MR, Monk BJ, Herrstedt J, Oza AM, Mahner S, Redondo A, Fabbro M, Ledermann JA, Lorusso D, Vergote I, Ben-Baruch NE, Marth C, Madry R, Christensen RD, Berek JS, Dorum A, Tinker AV, du Bois A, Gonzalez-Martin A, Follana P, Benigno B, Rosenberg P, Gilbert L, Rimel BJ, Buscema J, Balser JP, Agarwal S, Matulonis UA; ENGOT-OV16/NOVA Investigators. Niraparib Maintenance Therapy in Platinum-Sensitive, Recurrent Ovarian Cancer. N Engl J Med. 2016 Dec 1;375(22):2154-2164. doi: 10.1056/NEJMoa1611310. Epub 2016 Oct 7. PMID 27717299
- [Background] Romero I, Rubio MJ, Medina M, Matias-Guiu X, Santacana M, Schoenenberger JA, Guerra EM, Cortes A, Minig L, Coronado P, Cueva JF, Gomez L, Malfettone A, Sampayo M, Llombart-Cussac A, Poveda A. An olaparib window-of-opportunity trial in patients with early-stage endometrial carcinoma: POLEN study. Gynecol Oncol. 2020 Dec;159(3):721-731. doi: 10.1016/j.ygyno.2020.09.013. Epub 2020 Sep 26. PMID 32988624